CLINICAL TRIAL: NCT06348108
Title: A Phase Ib, Multi-center, Study of Talquetamab in Combination With Iberdomide and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Talquetamab in Combination With Iberdomide and Dexamethasone for Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Martin, MD (Other)
Collaborators: Janssen Research & Development, LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Thomas Martin, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 232514; NCI-2024-01992 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma; Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; iberdomide; Dexamethasone; Calcium Dobesilate; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Cohort: Dose Level (DL) 1 (Talquetamab, Iberdomide, Dexamethasone) - Starting Dose (Experimental): Participants receive 0.8 mg/kg Talquetamab (Tal) subcutaneously (SQ) over 1-3 minutes every 2 weeks (days 1 and 15 of each cycle), 0.75 mg Iberdomide orally (PO) once a day (QD) on days 1-21 of each 28-day cycle, and 20-40mg of Dexamethasone PO weekly, but may be continued at the discretion of the investigator. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also undergo bone marrow biopsy, skeletal x-ray, CT, Positron Emission Tomography (PET)/CT, or MRI, tissue and blood sample collection throughout the study.
  Interventions: Biological: Talquetamab; Drug: Iberdomide; Drug: Dexamethasone; Procedure: Bone Marrow Biopsy
- Dose Escalation Cohort: DL 2 (Talquetamab, Iberdomide, Dexamethasone) (Experimental): Participants receive 0.8 mg/kg Talquetamab (Tal) subcutaneously (SQ) over 1-3 minutes every 2 weeks (days 1 and 15 of each cycle), 1.0 mg Iberdomide orally (PO) once a day (QD) on days 1-21 of each 28-day cycle, and 20-40mg of Dexamethasone PO weekly, but may be continued at the discretion of the investigator. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Participants also undergo bone marrow biopsy, skeletal x-ray, CT, Positron Emission Tomography (PET)/CT, or MRI, tissue and blood sample collection throughout the study.
  Interventions: Biological: Talquetamab; Drug: Iberdomide; Drug: Dexamethasone; Procedure: Bone Marrow Biopsy
- Dose Expansion Cohort (Talquetamab, Iberdomide, Dexamethasone) (Experimental): Participants receive the recommended phase 2 dose of Iberdomide in combination with Talquetamab and 20-40mg of Dexamethasone which may be continued at the discretion of the investigator. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Participants also undergo bone marrow biopsy, imaging scans, tissue and blood sample collection throughout the study.
  Interventions: Biological: Talquetamab; Drug: Iberdomide; Drug: Dexamethasone; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Biological: Talquetamab — Given subcutaneously (SQ)
  Other Names: Anti-CD3/Anti-GPRC5D Bispecific Monoclonal Antibody JNJ-64407564; DuoBody Antibody JNJ-64407564
Drug: Iberdomide — Given orally (PO)
  Other Names: CELMoD; CC-220; 1323403-33-3
Drug: Dexamethasone — Given PO
  Other Names: Decadron; DexPak; Hemady
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy

SUMMARY:
This phase I trial will evaluate the safety, side effects, and best dose of talquetamab in combination with iberdomide and dexamethasone in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or has not responded to previous treatment (refractory). There is currently a significant unmet need for patients with relapsed or refractory multiple myeloma (RRMM) who are triple class refractory and have been exposed to B-cell maturation antibody (BCMA) targeted therapy. These patients currently have limited treatment options and poor survival. Talquetamab is an FDA approved drug that can bring T-cells to the myeloma cell, resulting in myeloma cell death. Iberdomide is an investigational drug and works by targeting and destroying proteins that help myeloma cancer cells to survive. Dexamethasone is a corticosteroid, is similar to a natural hormone produced by the adrenal glands to reduce inflammation (swelling, heat, redness, and pain) and is used to in helping to treat certain types of cancer including myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety of the combination of talquetamab (Tal), iberdomide (Iber) and dexamethasone (Dex) in patients with triple class exposed (TCE) RRMM. (Phase 1b-dose escalation (DE)).

II. To assess dose limiting toxicity (DLT) and determine the recommended phase 2 dose (RP2D) of the combination of Tal, Iber and Dex administered in 28-day cycles in patients with TCE RRMM. (Phase 1b-DE).

III. To further assess safety of RP2D of the combination of Tal, Iber and Dex administered in 28-day cycles in patients with TCE RRMM Len-refractory, and having received >= 2 prior lines of therapy. (Phase 1b-expansion (Exp)).

IV. To assess overall response rate (ORR) in patients with TCE RRMM, Len-refractory, and having received ≥ 2 prior lines of therapy. (Phase 1b-Exp).

SECONDARY OBJECTIVES:

I. To assess ORR, and to determine minimal residual disease (MRD) negative (-) rates in patients achieving ≥ very good partial remission (VGPR).

II. To assess toxicity (incidence of adverse events (AEs), serious AEs (SAEs), and treatment discontinuation due to toxicity) and safety (physical examination findings, vital signs, and clinical laboratory evaluations) in patients with RRMM.

III. Describe changes in health-related quality of life (HRQoL) using the European Organization for Research and Treatment of Cancer (C30) -Quality of Life questionnaire (QLQ) (EORTC-QLQ-C30), EORTC QLQ Oral Health 15 (OH-15) and EORTC QLQ-Multiple Myeloma Questionnaire (MY20)).

EXPLORATORY OBJECTIVES:

I. To assess serum cytokines levels with treatment of the combination of Tal, Iber and Dex and the predictive values of response, cytokine release syndrome (CRS) and other adverse events.

II. To assess changes in immune cells in blood and bone marrow with treatment of the combination of Tal, Iber and Dex.

III. To determine the efficacy of combination of Tal, Iber and Dex defined as Objective Response Rate (ORR) and achieving complete response (CR) and MRD (-) status and correlation between mass spectroscopy and bone marrow (BM) MRD assessments.

OUTLINE: This is a dose-escalation study of Iber followed by a dose-expansion study.

Participants receive Tal in cycle 1 then all 3 drugs will be given in combination in cycle 2 but may be continued at the discretion of the investigator. Cycles repeat every 28 days for as long as there is clinical benefit as determined by the Investigator. Study treatment will be discontinued if there is unacceptable toxicity, disease progression, withdrawal of consent by the participant, noncompliance with study requirements, intercurrent illness, or closure of the study by the Sponsor.

After completion of study treatment, patients are followed up at 30 days every 8 weeks for up to 3 years or until progression or initiation of subsequent therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Has a prior history of (h/o) MM (based on International Myeloma Working Group (IMWG) criteria) and now has evidence of relapsed or refractory MM. RRMM of progressive disease as defined by the IMWG 2006 and 2016 criteria (Kumar at al).
3. Specific criteria for dose escalation and dose expansion:

   1. Phase 1 dose escalation: patients will be required to have TCE RRMM (including a proteasome inhibitor (PI) (≥ 2 cycles or 2 months of treatment), an immunomodulatory drug (IMiD)) (≥ 2 cycles or 2 months of treatment) and a CD38 antibody (≥ 2 cycles or 2 months of treatment) after receiving ≥ 3 prior lines of therapy. Prior BCMA exposure is allowed. (Subjects with discontinued PI/IMiD/Cluster of differentiation 38 (CD38) therapy due to severe adverse event after < 2 months are allowed)
   2. Dose expansion cohort: RRMM patients will be lenalidomide refractory, TCE (exposed to IMiD, PI and CD38 antibody therapy (≥ 2 cycles or 2 months of treatment for each) and have received ≥ 2 prior lines of therapy. Prior BCMA targeted therapy is allowed, not required. (Subjects with discontinued PI/IMiD/CD38 therapy due to severe adverse event after < 2 months are allowed. Lenalidomide refractory is defined as having evidence of progressive disease on lenalidomide (≥ 10 mg or greater, ≥ 21 days/28) or within 60 days of stopping lenalidomide therapy.)
4. Has measurable disease defined as at least 1 of the following:

   1. Serum M-protein ≥ 0.5 g/dL (dose escalation) and 1.0 g/dL (dose expansion cohorts)
   2. Urine M-protein ≥ 200 mg/24 hours
   3. Serum free light chain (FLC) assay: involved FLC assay ≥ 10 mg/dL (≥ 100 mg/L) AND an abnormal serum FLC ratio (< 0.26 or > 1.65). (Can be used to fulfill the inclusion criteria of measurable disease in patients who do not have measurable disease by M-protein).
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Has adequate baseline organ function, as demonstrated by the following:

   1. Calculated creatinine clearance > 30 mL/min as assessed by the Cockcroft-Gault equation, Modification of Diet in Renal Disease (MDRD) equation (National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), 2015) or as assessed by 24-hour urine collection.
   2. Serum bilirubin ≤ 1.5 mg/dL, excluding Gilbert's.
   3. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × institutional upper limit normal (ULN).
   4. Total serum calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL) (treatment of hypercalcemia is allowed and patients may enroll if hypercalcemia returns to WNL with standard treatment).
7. Has adequate baseline hematologic function, as demonstrated by the following:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L (myeloid growth factors must not have been administered within 7 days (14 days for extended 1/2-life products).
   2. Hemoglobin ≥ 8 g/dL (red blood cell transfusions permitted provided the anemia is disease-related).
   3. Platelet count ≥ 100 x 10^9/L and no platelet transfusions during the 7 days before first dose (without transfusions). (Dose expansion cohorts will be allowed to have platelets counts ≥ 75 x 10^9/L with no platelet transfusions during the prior 7 days).
8. Must have at least 2 negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test result obtained prior to initiating therapy. The first test should be performed within 10-14 days and the second within 24 hours prior to initiating therapy if the patient is a female of childbearing potential (FCBP; defined as a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy or has not been naturally postmenopausal for at least 24 consecutive months).
9. Men and women of childbearing potential must agree to not donate sperm and eggs (ova and oocytes) throughout study therapy and for 3 months after the last treatment.
10. Men and women agree to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 3 months after the last treatment with study treatment.

    1. Women of childbearing potential must agree to 2 methods of reliable birth control simultaneously while receiving study treatment and until 100 days after last dose of study treatment: one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [oral, injectable, transdermal patches, vaginal rings or implants] or partner's vasectomy, and 1 additional effective contraceptive method (male latex or synthetic condom, diaphragm or cervical cap).
    2. Males must agree to always use a latex or synthetic condom during any sexual contact with females of reproductive potential.
11. All patients should be encouraged to be fully vaccinated prior to initiation of therapy including being up-to-date on vaccines against pneumococcus, yearly influenza, Coronavirus disease (COVID) booster(s), and any age appropriate vaccine. Live attenuated vaccines are not allowed while on study treatment or within 4 weeks of starting treatment.
12. Has provided signed informed consent before initiation of any study-specific procedures or treatment.
13. Must agree to, and be capable of, adhering to the study visit schedule and other protocol requirements, including follow-up for overall survival.

Exclusion Criteria:

1. Has persistent clinically significant toxicities (grade ≥ 2; per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) from previous anticancer therapy (excluding alopecia which is permitted and excluding grades 2 and 3 laboratory abnormalities (including hematologic abnormalities) if participants are not associated with symptoms, are not considered clinically significant by the investigator, and can be managed with available medical therapies.
2. Has NCI CTCAE grade ≥ 3 peripheral neuropathy from any etiology or grade ≥ 2 peripheral neuropathy with pain.
3. Has received treatment with cytotoxic (alkylators) within 3 weeks, biologic (IMiDs/PIs) within 2 weeks, targeted therapies (monoclonal antibodies) within 4 weeks, chimeric antigen receptor (CAR) T-cell (CAR-T)or autologous stem cell transplant therapy within 3 months or any novel therapy within 5- 1/2 lives of therapy.
4. Has had radiation therapy within 14 days of first dose of study therapy, unless less than 5% marrow exposure, then no limit.
5. Has had any prior GPRC5D targeted bispecific antibody therapy or GPRC5D CAR-T therapy or has had previous treatment with Iber.
6. Has any active or uncontrolled infection including any viral, bacterial or fungal infection; and/or HIV, active hepatitis (Hep) C and active Hep B (hepatitis B (HB) surface antigen (HBsAg) (+), HB core antigen (HBcAb) (+) or (+) Hep B deoxyribonucleic acid (DNA) by polymerase chain reaction (pcr), Hep C ribonucleic acid (RNA) (+) by pcr. Patients who have received Intravenous immunoglobulin therapy (IVIG) replacement therapy may have (+) HBcAb results from the IVIG therapy. These patients can enroll if Hep B DNA by pcr test is negative. These patients need to be on antiviral therapy and be monitored for hepatitis B virus (HBV) DNA throughout study therapy per local guidelines and as clinically indicated.
7. Has an additional active malignancy that may confound the assessment of the study endpoints. If the patient has a past cancer history (active malignancy within 2 years before study entry) with substantial potential for recurrence, this must be discussed with the sponsor/investigator before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: nonmelanoma skin cancer and carcinoma in situ (including transitional cell carcinoma, cervical cancer, anal carcinoma, ductal carcinoma in situ (DCIS) and melanoma in situ), any cancer resected with curative intent, low-grade cancer not requiring therapy.
8. Is pregnant or breast feeding.
9. Has clinically significant cardiovascular disease including, albeit not limited to:

   1. Uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure
   2. Uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months before study entry
   3. Uncontrolled hypertension or clinically significant arrhythmias not controlled by medication.
10. Has active POEMS (polyneuropathy, organomegaly, endocrinopathy/edema, monoclonal-protein, skin syndrome), amyloid light (AL) amyloidosis, primary plasma cell leukemia or active central nervous system (CNS) or parenchymal/leptomeningeal myeloma.
11. Has uncontrolled, clinically significant organ dysfunction that in the opinion of the investigator would put the patient at significant risk for toxicity from study therapy.
12. Has recent major surgery within 4 weeks or significant gastrointestinal (GI) disease that would interfere with GI absorption of oral medications.
13. Has a condition, including autoimmune disease, requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days before study therapy administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
14. Has received treatment with allogeneic stem cell transplant within 6 months before the first dose of study treatment and if > 6 months from allogeneic stem cell transplantation (alloSCT) must be off all immunosuppression and without evidence of active graft-versus-host disease (GVHD).
15. Uncontrolled epilepsy or new/recent seizure activity within 6 months of study entry.
16. Live vaccine administered within 4 weeks prior to study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants reporting treatment-emergent adverse events (AEs) (Dose Escalation Cohorts) | Up to 1 cycle (Cycles are 28 days in length)
  Safety will be evaluated for the population of participants who received at least one dose of study drug. Treatment-emergent AEs will be graded by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Proportion of participants experiencing Dose-Limiting Toxicity (DLTs) (Dose Escalation Cohorts) | Up to 1 cycle (Cycles are 28 days in length)
  Maximum tolerated dose (MTD) will be defined as the highest dose at which no more than one instance of DLT is observed among 6 participants treated.
Recommended phase 2 dose (RP2D) (Dose Escalation Cohorts) | Up to 1 cycle (Cycles are 28 days in length)
  RP2D will be defined as the MTD to be evaluated in the expansion cohort based on safety and preliminary activity of at least 2 dose levels (6 patients treated/dose level).
Proportion of participants experiencing Dose-Limiting Toxicity (DLTs) (Dose Expansion Cohort) | Up to 3 years
  The frequency, type, and severity (grade) of each DLT will be reported
Objective response rate (ORR) (Dose Expansion Cohort) | Up to 3 years
  ORR will be defined as all responses greater than or equal to a partial response (PR) (i.e., PR, very good partial response (VGPR), complete response (CR), or stringent complete response (sCR) per International Myeloma Working Group (IMWG) definition). Under Simon's two-stage design, final efficacy evaluation for the primary endpoint will calculate the uniformly minimum variance unbiased estimator, p-value and 95% CI for the response rates.

SECONDARY OUTCOMES:
Objective response rate (ORR) (Dose Escalation Cohorts) | Up to 3 years
  ORR will be defined as all responses greater than or equal to a partial response (i.e., PR, VGPR, CR, or sCR per IMWG definition). Will be summarized using frequency and percentage, along with 95% CIs.
Number of participants achieving VGPR or CR and MRD (negative (-)) response | Up to 3 years
  MRD will be defined as achieving ≥ VGPR and MRD (-) response will be defined as having < 1 multiple myeloma clone per 100,000 bone marrow cells (10-5) by next-generation sequencing (NGS) (clono sequence (seq); 10-5). Will be reported for the entire population and for those treated at the MTD.
Proportion of participants with treatment-related adverse events | Up to 3 years
  Toxicity will be measured by CTCAE version 5.0; cytokine release syndrome and immune effector cell-associated neurotoxicity syndrome (ICANS) will be assessed according to the American Society for Transplantation and Cellular Therapy guidelines; neurological treatment-emergent adverse events that are not assessed as ICANS should be graded per CTCAE version 5.0 and managed by per institutional guidelines.
Changes in scores on the European Organization for Research and Treatment of Cancer - Quality of Life questionnaire (EORTC-QLQ-C30) over time | Up to 3 years
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning.
Changes in scores on the EORTC QLQ- Multiple Myeloma Questionnaire (EORTC-QLQ-M20) over time | Up to 3 years
  The EORTC QLQ-MY20 is a 20-item questionnaire that is designed to measure the quality of life of people with multiple myeloma. Scores consists of responses to items addressing multiple myeloma-related symptoms and quality of life issues with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Calfornia, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No